CLINICAL TRIAL: NCT02519192
Title: The Role of VAC Therapy Devices in Promoting Closure of Enterocutaneous Fistulae: A Randomized Controlled Trial
Brief Title: The Role of VAC Therapy Devices in Promoting Closure of Enterocutaneous Fistulae
Acronym: ECF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research personal no longer available
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-2133
Record Dates: First submitted 2015-07-28; First posted 2015-08-10 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Fistulae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAC Arm, Vac sponge irrigations (Experimental): For patients who fall under the VAC arm, a physician will do the initial placement of the wound VAC (V.A.C.Ulta™ Negative Pressure Wound Therapy System) at the patient's bedside. An information sheet will be provided to the patient, and the patient will be taught how to irrigate the sponge system independently. While inpatient, nursing will perform VAC sponge irrigation.
  Interventions: Device: V.A.C.Ulta™ Negative Pressure Wound Therapy System; Procedure: Vac sponge irrigations
- NonVac, ostomy bag, wet to dry dressings (Active Comparator): For patients who fall under the non-VAC arm, a physician or wound care nurse will perform the initial application of the ostomy bag or wet to dry dressing change. An information sheet will be provided to the patient. While inpatient, members from the nursing or physician team will perform ostomy bag application and ostomy dressing changes.
  Interventions: Procedure: ostomy bag; Procedure: wet to dry dressings

INTERVENTIONS:
Device: V.A.C.Ulta™ Negative Pressure Wound Therapy System — VAC Arm will consist of a group of patients assigned to VAC negative pressure therapy with regular sponge irrigation with normal saline (the V.A.C.Ulta™ Negative Pressure Wound Therapy System) .
  Arms: VAC Arm, Vac sponge irrigations
Procedure: Vac sponge irrigations — VAC Arm will consist of a group of patients assigned to VAC negative pressure therapy with regular sponge irrigation with normal saline (the V.A.C.Ulta™ Negative Pressure Wound Therapy System) .
  Arms: VAC Arm, Vac sponge irrigations
Procedure: ostomy bag — Non Vac Arm will receive ostomy bag applications.
  Arms: NonVac, ostomy bag, wet to dry dressings
Procedure: wet to dry dressings — Non Vac arm will receive wet to dry dressing changes.
  Arms: NonVac, ostomy bag, wet to dry dressings

SUMMARY:
This study hopes to determine if a negative pressure dressing is superior to a traditional dressing for speeding fistula closure after laparotomy. This study has a broad variety of implications. Patient safety is a paramount concern: Investigators hope to identify a superior method of wound management which minimizes risk for skin breakdown, sepsis, and morbidity. In addition, patient satisfaction would be improved with a method for faster wound healing. Finally,implications exist in the realm of a cost-benefit analysis, for example, although the VAC method is more costly, it may save money if it speeds healing and prevents the need for reoperation. Alternatively, if the VAC method is not shown to be beneficial, physicians can avoid using a more costly device with no proven benefit.

DETAILED DESCRIPTION:
Investigators are planning a superiority trial to show that VAC use speeds the closure of enterocutaneous fistulae over routine gravity drainage. The investigators' design is a randomized controlled trial with two arms. One of the arms (non-VAC) will include patients assigned to a system of ECFoutput management which does not involve negative pressure (for example, an ostomy bag placed over the fistula, wet to dry dressing changes, etc..), and the second arm (VAC) will consist of a group of patients assigned to VAC negative pressure therapy with regular sponge irrigation with normal saline (the V.A.C.Ulta™ Negative Pressure Wound Therapy System) .

The fistula vac is made from standard sponge supplies and negative pressure suction devices. Initial placement will be by the bedside physician in the intensive care unit, the ward, or in the clinic. The patient will be taught basic wound care, and as is typical for those outpatients with wound VACs, a home nursing aide will be arranged. Those randomized to no VAC therapy will have ostomy bags or wet to dry dressings placed on the skin with no negative pressure applied. Again, initial application will be performed by the bedside physician or a wound care nurse. The patient will be taught wound care, with assistance provided as necessary.

Once a fistula is noted to have closed (effluent = 0cc/day) the dressings or VAC will be discontinued, and the date of fistula closure noted.

ELIGIBILITY:
Inclusion Criteria:

* post-laparotomy patient developing a new enterocutaneous fistula

Exclusion Criteria:

* patient with a prior history of abdominal radiation
* patient with a distal obstruction, any entero-atmospheric fistula, or any patient with a history of intra-abdominal or metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
primary endpoint of time to fistula closure | Expected average of 6-8 weeks
  Study subjects will be followed until closure of the enterocutaneous fistula, an expected average of 6-8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD MPH, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No